CLINICAL TRIAL: NCT01528826
Title: A Prospective Phase II Trial of Vinorelbine Plus Oxaliplatin in Pretreated Metastatic Triple-negative Breast Cancer
Brief Title: Salvage Chemotherapy of Vinorelbine Plus Oxaliplatin in Metastatic Triple-negative Breast Cancer:a Prospective Trial
Acronym: NVBOX
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, yanfei Liu, principal investigator, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NVBOX
Record Dates: First submitted 2012-01-29; First posted 2012-02-08 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Breast Cancer
Keywords: metastatic triple-negative breast cancer; vinorebine; oxaliplatin
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — Vinorelbine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NVBOX regimen (Experimental): Vinorelbine plus oxaliplatin
  Interventions: Drug: vinorelbine plus oxaliplatin

INTERVENTIONS:
Drug: vinorelbine plus oxaliplatin — Vinorelbine 30mg/m2 IVGTT D1 Oxaliplatin 90mg/m2 IVGTT D1; every 2 weeks

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of vinorelbine plus oxaliplatin in pretreated metastatic triple-negative breast cancer.

DETAILED DESCRIPTION:
Triple-negative breast cancer is associated with less treatment choices and shorter overall survival. Both vinorebine and oxaliplatin are effective in metastatic breast cancer. The investigators designed this trial to evaluate the combination of these two drugs in pretreated metastatic triple-negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Females with age between 18 and 70 years old
2. ECOG performance between 0-2
3. Life expectancy more than 3 months
4. Histological proven unresectable recurrent or advanced breast cancer
5. Triple-negative for estrogen receptor (ER), progestogen receptor (PR), and human epithelial receptor-2 (HER2) by immunohistochemistry (IHC) test. For patients with ER negative, PR negative, Her2 two plus, a negative Her2 gene amplification should be verified with FISH test. Her2 one plus may consider FISH verification.
6. No more than 2 chemotherapy for metastatic breast cancer.
7. At least one measurable disease according to the response evaluation criteria in solid tumor (RECIST1.1)
8. No anticancer therapy within 4 weeks
9. No neuropathy more than grade I
10. Adequate hematologic, hepatic, and renal function,No serious medical history of heart, lung, liver and kidney
11. Provision of written informed consent prior to any study specific procedures

Exclusion Criteria:

1. Pregnant or lactating women (female patients of child-bearing potential must have a negative serum pregnancy test within 14 days of first day of drug dosing, or, if positive, a pregnancy ruled out by ultrasound)
2. Women of child-bearing potential, unwilling to use adequate contraceptive protection during the course of the study
3. Treatment with an investigational product within 4 weeks before the first treatment
4. Symptomatic central nervous system metastases
5. Other active malignancies (including other hematologic malignancies) or other malignancies, except for cured nonmelanoma skin cancer or cervical intraepithelial neoplasia.
6. Patient having a history of clinically significant cardiovascular, hepatic, respiratory or renal diseases, clinically significant hematological and endocrinal abnormalities, clinically significant neurological or psychiatric conditions
7. Uncontrolled serious infection
8. Previous administration of vinorelbine
9. Patients with bad compliance

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2011-12; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
progression free survival | 6 weeks

SECONDARY OUTCOMES:
overall response rate | 6 weeks
overall survival | 6 weeks
Safety and Tolerability | 6 weeks
  Number of Participants with Adverse Events, Degree of Adverse Events according to CTC4.0
genetic polymorphisms | 6 weeks
  To evaluate the relationship of genetic polymorphisms and efficacy.

CONTACTS AND LOCATIONS:
Overall Officials: Zhonghua Wang, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Cancer Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Zhang J, Wang L, Wang Z, Hu X, Wang B, Cao J, Lv F, Zhen C, Zhang S, Shao Z. A phase II trial of biweekly vinorelbine and oxaliplatin in second- or third-line metastatic triple-negative breast cancer. Cancer Biol Ther. 2015;16(2):225-32. doi: 10.4161/15384047.2014.986973. PMID 25648299